CLINICAL TRIAL: NCT04405297
Title: A Disease-based Treatment Study for Diagnosed Osteoarthritis Utilizing Adipose-derived Regenerative Cells
Status: Terminated | Type: Observational
Why Stopped: The sponsor decided to close the study early due to low patient enrollment and the sponsor no longer pursuing stem cell therapy treatment.
Sponsor: Sanford Health (Other)
Responsible Party: Sponsor
Other Study IDs: ENDURE
Record Dates: First submitted 2020-05-08; First posted 2020-05-28 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Knee Osteoarthritis; Hip Osteoarthritis; Ankle Osteoarthritis; Shoulder Osteoarthritis; Wrist Osteoarthritis
Keywords: Stem Cells; Adipose-derived regenerative cells; Osteoarthritis; Adipose-derived stem cells; Arthritis; Joint Diseases
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Osteoarthritis; Arthritis; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — After completion of the product release criteria testing, a small amount of the sample will be processed and stored for future research. These retained samples will be used for future research. Future research results will not be returned to the study participants or investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (5):
- Hip Osteoarthritis: Subjects will receive autologous adipose-derived regenerative stem cells into their affected hip joint.
  Interventions: Device: Adipose-derived regenerative cells
- Knee Osteoarthritis: Subjects will receive autologous adipose-derived regenerative stem cells into their affected knee joint.
  Interventions: Device: Adipose-derived regenerative cells
- Ankle Osteoarthritis: Subjects will receive autologous adipose-derived regenerative stem cells into their affected ankle joint.
  Interventions: Device: Adipose-derived regenerative cells
- Shoulder Osteoarthritis: Subjects will receive autologous adipose-derived regenerative stem cells into their affected shoulder joint.
  Interventions: Device: Adipose-derived regenerative cells
- Wrist Osteoarthritis: Subjects will receive autologous adipose-derived regenerative stem cells into their affected wrist joint.
  Interventions: Device: Adipose-derived regenerative cells

INTERVENTIONS:
Device: Adipose-derived regenerative cells — Adipose-derived regenerative cells will be obtained from a small-volume lipoaspirate procedure. The lipoaspirate will then be enzymatically digested to produce a stromal vascular fraction (SVF) that will be injected into the targeted joint.

SUMMARY:
This is a prospective, multi-location safety and effectiveness study, and data registry of autologous adult ADRCs generated by the Transpose® RT System in subjects with OA in the shoulder, wrist, knee, hip, or ankle.

DETAILED DESCRIPTION:
Subjects who have signed informed consent and Health Insurance Portability and Accountability Act (HIPPA) authorization, and are determined to meet all inclusion criteria and no exclusion criteria will be enrolled in this study and receive the ADRC treatment.

The subject will have an injection procedure (ADRC treatment) For this study, a licensed physician trained in liposuction must perform the syringe liposuction procedure. The licensed physician who performs the lipoplasty may be the Investigator or a non-Investigator physician (e.g., a plastic surgeon) who is trained on the study protocol.

All subjects will undergo a minor syringe liposuction procedure to acquire approximately 100 mL of lipoaspirate for preparation of ADRC using the Transpose® RT System. The removed tissue is processed to extract a cell suspension (the cell product). Once the cell product has been obtained, tested, and found to conform to release criteria, the subject will be treated with the ADRCs.

ELIGIBILITY:
All Cohorts:

To be eligible to participate in this study, a subject must meet all the following criteria.

Inclusion Criteria-ALL Cohorts:

1. Men and women age 18 or older
2. Clinical and radiographic diagnosis of OA in one of the following areas: Ankle, Hip, Knee, Shoulder, or Wrist
3. Continued OA pain in the targeted joint despite conservative measures (per treating provider's discretion)
4. Average daily VAS Pain Score ≥3
5. Understand and provide written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization prior to initiation of any study-specific procedures
6. On physical exam. subject appears to have adequate adipose tissue for liposuction
7. Subject must also meet additional inclusion criteria specific to the targeted joint cohort

Ankle Cohort:

1. Currently Kellgren-Lawrence Grade II, III or IV in the ankle based on X-ray (weight-bearing mortise views with 20⁰ internal rotation)
2. Ankle pain for at least 6 months, despite conservative treatment or inability to tolerate the side effects of medications
3. Normal activity level, not bedridden or confined to a wheelchair, able to walk 30 meters without the aid of a walker, crutches or cane

Hip Cohort:

1. Hip OA diagnosed on x-ray and/or Magnetic Resonance Imaging (MRI) (Tӧnnis grade 1, 2, or 3)

Knee Cohort:

1. Kellgren-Lawrence system of Grade II, III, or IV
2. Subject may have concomitant patellofemoral but they must have stage II or higher generalized knee OA

Shoulder Cohort:

1. Grades 1, 2 or 3 OA in the index glenohumeral joint based on the Samilson-Prieto classification system as confirmed by X-ray (axillary view and true anterior-posterior view)
2. Subjects who have failed standard non-surgical management of their shoulder arthritis who would benefit from a shoulder arthroplasty. Failed medical management will be defined as persistent pain and disability despite adequate standard non-operative management for 6 months. Medical management will be defined as:

   1. The use of drugs including analgesics and non-steroidal anti-inflammatory drugs
   2. Activity modification

Wrist Cohort:

1. Clinical symptoms consistent with wrist OA

Exclusion Criteria- ALL Cohorts:

1. Subject cannot meet any of the exclusion criteria listed of the targeted joint cohort
2. Viscosupplementation within 6 months of screening in the targeted joint
3. Other Biologic Injection (Platelet Rich Plasma (PRP) or stem cell) within 6 months in the targeted joint
4. Surgery in the targeted joint within the past 6 months (either open or scope)
5. Planned/anticipated surgery of the targeted joint during study participation
6. Systemic or intra-articular injection of corticosteroids in any joint within 3 months before screening (re-screening allowed once this criteria is met)
7. Females of childbearing age who have not used or do not plan to use acceptable birth control measures, for the duration of the study. Oral, injected or implanted hormonal contraceptive, barrier methods (condom or diaphragm with spermicide), intrauterine device, surgical sterilization, transdermal delivery, congenital sterility or sexual abstinence are considered acceptable forms of birth control. If sexually active, the subject must have been using one of the accepted birth control methods at least one month prior to study entry.
8. Part of a vulnerable population per Office for Human Research Protections (OHRP) definition (pregnant women and breast-feeding women, cognitively impaired, prisoners, etc.)
9. Unwilling to discontinue the use of Non-Steroidal Anti-Inflammatory (NSAID)s for 7 calendar days prior to the procedure
10. Unwilling to discontinue NSAIDS for 5 calendar days after procedure
11. Insufficient amount of subcutaneous tissue to allow recovery of at least 100mL of lipoaspirate
12. Diagnosed musculoskeletal cancer or any diagnosed cancer, other than musculoskeletal if not on long term remission (e.g. at least 5 years or negative biopsy at last exam), except basal cell carcinoma
13. Have received chronic (more than 7 consecutive days) treatment with systemic corticosteroids at a dose equivalent to prednisone ≥ 10 mg/day within 14 days prior to an injection procedure.
14. Subject is currently participating in another clinical trial that has not yet completed its primary endpoint. (Nonintervention observational studies are not exclusionary.)
15. History of, or ongoing, autoimmune disorder that requires treatment with an immunosuppressive medication
16. Subjects who have a documented history or presence of inflammatory arthritis, rheumatoid arthritis, and sepsis in the treatment site
17. History of bleeding disorders or inflammatory joint disease
18. Inability to hold anti-platelet therapy according to treating provider prior to procedure
19. Any medical condition that could preclude participation in the study in the opinion of the investigator
20. Active workers' compensation case in progress with the targeted joint
21. Daily opioid use for the 3 months prior to screening or anticipated daily use while participating on study
22. Psychiatric disorder that may prevent participation in the study in the opinion of the investigators
23. A positive screen for human immunodeficiency virus (HIV) by antibodies or nucleic acid test
24. Has a known active Hepatitis B (e.g. HBsAg reactive) or Hepatitis C (e.g. HCV RNA [qualitative] is detected)
25. Allergy to sodium citrate of any "caine" type of local anesthetic
26. Hemoglobin less than 10g/dL at the time of screening
27. Leukocytes <3,000/µL; neutrophils <1,500/µL; lymphocytes <800/µL; platelets <100,000/µL at the time of screening
28. Subjects with a known diagnosis of osteoporosis
29. Diagnosis of liver disease as defined by alanine aminotransferase (ALT) >2x the upper limit of age-determined normal (ULN) or total bilirubin > 1.5x ULN

Ankle Cohort:

1. Lower leg trauma in a location other than within the ankle
2. Arthroscopy or open surgery of the ankle joint within 6 months of screening.
3. Extreme obesity, as defined by National Institutes of Health (NIH) Clinical Guidelines Body Mass Index (BMI > 40)
4. Any condition other than OA of the ankle joint which, in the opinion of the investigator, affects their ability to ambulate to a sufficient degree to interfere with the assessment of the safety and treatment effects of the study injection.

Hip Cohort:

1. Evidence of hip dysplasia (centre edge angle less than 20⁰)
2. Previous fracture trauma to the affected hip requiring medical or surgical treatment
3. Severe acetabular deformities (e.g. acetabular protrusion, coxa profunda, circumferential labral ossification)
4. Infections or skin diseases at target hip joint
5. Significant medical co-morbidities (requiring daily assistance for activities of daily living)
6. Any clinically significant or symptomatic vascular or neurologic disorder of the lower extremities
7. Extreme obesity, as defined by NIH Clinical Guidelines Body Mass Index (BMI>40)
8. Femoral head deformity (perthes or AVN)

Knee Cohort:

1. Extreme obesity, as defined by NIH Clinical Guidelines Body Mass Index (BMI>40)
2. Clinically apparent tense effusion of the targeted knee
3. Significant valgus/varus deformities (+/- 10⁰)

Shoulder Cohort:

1. Walch B2 glenoid with greater than 10⁰ of retroversion
2. Active joint or systemic infection
3. Rotator cuff arthropathy
4. Significant muscle paralysis
5. Charcot's arthropathy

Wrist Cohort:

1. Subjects who have a documented diagnosis of active carpal tunnel syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The focus of this study is to investigate the therapeutic benefit of autologous ADRCs in patients with OA in various joints. The ENDURE study allows subjects at Sanford Health and in the United States access to adipose-derived regenerative cells while reviewing safety for subjects with knee, shoulder, hip, ankle and wrist OA, using a more pragmatic and standard clinical approach.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Safety as indicated by incidence (%) of unanticipated AEs. All AEs and SAEs will be graded on severity by the Investigator using the National Institutes of Health Common Terminology Criteria for Adverse Events (NIH CTCAE). | Up to 2 years
  A one-sided binomial test will be used with a significance level of 0.05 to test whether safety was significantly lower than 20%. Each cohort will be analyzed independently.
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the knee using PROMIS 10 Global health | Through study completion, up to 3 years
  The PROMIS® is a set of participant-centered measures that evaluates and monitors the physical, mental, and social health in adults. Although unknown in osteoarthritis, the PROMIS® 10 Global Heath Survey was developed by the National Institute of Health and validated across a variety of chronic conditions. Each efficacy measure will be analyzed separately while accounting for potential confounding factors in the model such as age, sex, BMI, severity of OA diagnosis, smoking status, and past treatments in targeted joint. The Bonferroni adjustment for multiple testing correction will be used within each cohort. The PROMIS Global-10 is a 10-item patient-reported questionnaire utilizing as 5-point Global Physical Health Score scale ranging from 5="Excellent/Completely" to 1="Poor/Not at all" and a 5-point Global Mental Health scale ranging from 5="Never/None" to 1="Always/Very Severe", as well as a single 11-point question scale from 0="No Pain" to 10="Worst Pain Imaginable".
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the knee using SF-12v2 | Through study completion, up to 3 years
  The SF-12v2 is a generic health outcome measurement widely used in chronic illness and chronic pain conditions. The SF-12v2 is a shorter tool that requires less patient and provider effort. Validity and feasibility have been reviewed with demonstration for significance in non-cancer pain patients.Each efficacy measure will be analyzed separately while accounting for potential confounding factors in the model such as age, sex, BMI, severity of OA diagnosis, smoking status, and past treatments in targeted joint. The Bonferroni adjustment for multiple testing correction will be used within each cohort. SF-12v2 patient-reported questionnaire is utilizes a 5-point scale ranging from "Excellent"/"All of the time" to "None of the time"/"Poor" for both physical and mental questions as well as a 3-point score ranging from "Yes, limited a lot" to "No, not limited at all" for two physical questions.
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the knee using the Visual Analog Pain Scale (VAS-Pain) | Through study completion, up to 3 years
  A VAS instrument measures a characteristic that spans a continuum, cannot be precisely or optimally measured by or would lack sensitivity in distinguishing subtle changes on an ordinal scale. Pain intensity is a characteristic that is commonly measured in this manner. A 100-mm VAS will be administered to assess the subject's experience of joint pain intensity. Each efficacy measure will be analyzed separately while accounting for potential confounding factors in the model such as age, sex, BMI, severity of OA diagnosis, smoking status, and past treatments in targeted joint. The Bonferroni adjustment for multiple testing correction will be used within each cohort. The visual analog scale (VAS) patient-reported questionnaire is a subjective measure for acute and chronic pain utilizing a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain".
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the knee using the Knee Osteoarthritis Outcome Score (KOOS) | Through study completion, up to 3 years
  The Knee injury and Osteoarthritis Outcome Score (KOOS) is a valid, reliable, and responsive outcome measure in total joint replacement (E. T.-L. Roos 2003). KOOS is a self-administered questionnaire that assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life. Each efficacy measure will be analyzed separately while accounting for potential confounding factors in the model such as age, sex, BMI, severity of OA diagnosis, smoking status, and past treatments in targeted joint. The Bonferroni adjustment for multiple testing correction will be used within each cohort. The KOOS's patient-reported questionnaire utilizes 5-point Likert scale, options scored from 0 (No problems) to 4 (Extreme problems).
Efficacy outcomes include changes in the range of motion of the knee (ROM) measurements for the knee | Through study completion, up to 3 years
  Ranges include:
  0-140 degrees flexion 0 degrees extension
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the shoulder using PROMIS 10 Global health | Through study completion, up to 3 years
  The PROMIS® is a set of participant-centered measures that evaluates and monitors the physical, mental, and social health in adults. Although unknown in osteoarthritis, the PROMIS® 10 Global Heath Survey was developed by the National Institute of Health and validated across a variety of chronic conditions. Each efficacy measure will be analyzed separately while accounting for potential confounding factors in the model such as age, sex, BMI, severity of OA diagnosis, smoking status, and past treatments in targeted joint. The Bonferroni adjustment for multiple testing correction will be used within each cohort. The PROMIS Global-10 is a 10-item patient-reported questionnaire utilizing as 5-point Global Physical Health Score scale ranging from 5="Excellent/Completely" to 1="Poor/Not at all" and a 5-point Global Mental Health scale ranging from 5="Never/None" to 1="Always/Very Severe", as well as a single 11-point question scale from 0="No Pain" to 10="Worst Pain Imaginable".
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the shoulder using SF-12v2 | Through study completion, up to 3 years
  The SF-12v2 is a generic health outcome measurement widely used in chronic illness and chronic pain conditions. The SF-12v2 is a shorter tool that requires less patient and provider effort. Validity and feasibility have been reviewed with demonstration for significance in non-cancer pain patients. Each efficacy measure will be analyzed separately while accounting for potential confounding factors in the model such as age, sex, BMI, severity of OA diagnosis, smoking status, and past treatments in targeted joint. The Bonferroni adjustment for multiple testing correction will be used within each cohort. SF-12v2 patient-reported questionnaire is utilizes a 5-point scale ranging from "Excellent"/"All of the time" to "None of the time"/"Poor" for both physical and mental questions as well as a 3-point score ranging from "Yes, limited a lot" to "No, not limited at all" for two physical questions.
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the shoulder using the Visual Analog Pain Scale (VAS-Pain) | Through study completion, up to 3 years
  A VAS instrument measures a characteristic that spans a continuum, cannot be precisely or optimally measured by or would lack sensitivity in distinguishing subtle changes on an ordinal scale. Pain intensity is a characteristic that is commonly measured in this manner. A 100-mm VAS will be administered to assess the subject's experience of joint pain intensity. The visual analog scale (VAS) patient-reported questionnaire is a subjective measure for acute and chronic pain utilizing a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain".
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the shoulder using American Surgeon and Elbow Surgeon (ASES) measure | Through study completion, up to 3 years
  The ASES is a 100-point scale that consists of questions related to pain and activities of daily living. It is comprised of patient self-evaluation section and a physician assessment section.The activities of daily living questionnaire are marked on a four-point ordinal scale that can be converted to a cumulative activities of daily living index. The physician assessment section includes demographic information and assess range of motion, specific physical signs, strength and stability. A shoulder score can be derived from the visual analogue scale score for pain (50%) and the cumulative activities of daily living score (50%). The ASES is a 17-item patient-reported questionnaire utilizing a 10-point pain scale ranging from 0="No pain at all" to 10="Pain as bad as it can be" and a 4-point activities of daily living scale ranging from 0="Unable to do" to 3="Normal"
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the shoulder using the Oxford Shoulder Score | Through study completion, up to 3 years
  The Oxford Shoulder Score (OSS) is validated patient-reported outcome providing researchers and clinicians with a quantitative measure of a patient's response after a surgical and non-surgical shoulder intervention. Developed by the Department of Public Heath in the United Kingdom, the OSS is a 12-item tool used to review patient's pain and function, and is widely utilized in clinical trials. The Oxford Shoulder Score (OSS) is a 12-item patient-reported questionnaire utilizing as a 5-point Likert scale ranging from "None"/No trouble at all" to "Unbearable"/"Impossible to do".
Efficacy outcomes include changes in the range of motion of the shoulder (ROM) | Through study completion, up to 3 years
  Ranges include:
  0-180 degrees forward flexion 0-150 degrees abduction 30 degrees adduction 70-90 degrees internal rotation 0-90 degrees external rotation
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the wrist using PROMIS 10 Global health | Through study completion, up to 3 years
  The PROMIS® is a set of participant-centered measures that evaluates and monitors the physical, mental, and social health in adults. Although unknown in osteoarthritis, the PROMIS® 10 Global Heath Survey was developed by the National Institute of Health and validated across a variety of chronic conditions. Each efficacy measure will be analyzed separately while accounting for potential confounding factors in the model such as age, sex, BMI, severity of OA diagnosis, smoking status, and past treatments in targeted joint. The Bonferroni adjustment for multiple testing correction will be used within each cohort. The PROMIS Global-10 is a 10-item patient-reported questionnaire utilizing as 5-point Global Physical Health Score scale ranging from 5="Excellent/Completely" to 1="Poor/Not at all" and a 5-point Global Mental Health scale ranging from 5="Never/None" to 1="Always/Very Severe", as well as a single 11-point question scale from 0="No Pain" to 10="Worst Pain Imaginable".
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the wrist using SF-12v2 | Through study completion, up to 3 years
  The SF-12v2 is a generic health outcome measurement widely used in chronic illness and chronic pain conditions. The SF-12v2 is a shorter tool that requires less patient and provider effort. Validity and feasibility have been reviewed with demonstration for significance in non-cancer pain patients. Each efficacy measure will be analyzed separately while accounting for potential confounding factors in the model such as age, sex, BMI, severity of OA diagnosis, smoking status, and past treatments in targeted joint. The Bonferroni adjustment for multiple testing correction will be used within each cohort. SF-12v2 patient-reported questionnaire is utilizes a 5-point scale ranging from "Excellent"/"All of the time" to "None of the time"/"Poor" for both physical and mental questions as well as a 3-point score ranging from "Yes, limited a lot" to "No, not limited at all" for two physical questions.
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the wrist using the Pain Score Analog Scale (VAS-Pain) | Through study completion, up to 3 years
  A VAS instrument measures a characteristic that spans a continuum, cannot be precisely or optimally measured by or would lack sensitivity in distinguishing subtle changes on an ordinal scale. Pain intensity is a characteristic that is commonly measured in this manner. A 100-mm VAS will be administered to assess the subject's experience of joint pain intensity. Each efficacy measure will be analyzed separately while accounting for potential confounding factors in the model such as age, sex, BMI, severity of OA diagnosis, smoking status, and past treatments in targeted joint. The Bonferroni adjustment for multiple testing correction will be used within each cohort.
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the wrist using the Quick-Dash | Through study completion, up to 3 years
  The subject will complete the QuickDASH by scoring each item of the questionnaire with scores between 1 (no difficulty at all) and 5 (unable to do), with higher scores indicating greater disability (Hudak 1996, Kennedy 2011). The QuickDASH questionnaire is considered complete when 10 of the total 11 items are answered. The QuickDASH is an 11 item patient-reported questionnaire utilizing as a 5-point Likert scale ranging from 1="No difficulty"/"None" to 5="Unable to perform"/"Extreme".
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the wrist using PROMIS-Upper Extremity | Through study completion, up to 3 years
  The subject will complete the PROMIS self-report without help from anyone else. The respondents will be given the optimal time needed to capture the most relevant perspective and complete data (e.g., before/after clinician visit or in between visits). All results will be recorded and analyzed in accordance with standard practice. Each efficacy measure will be analyzed separately while accounting for potential confounding factors in the model such as age, sex, BMI, severity of OA diagnosis, smoking status, and past treatments in targeted joint. The Bonferroni adjustment for multiple testing correction will be used within each cohort.PROMIS- Upper Extremity is a 7-item patient-reported questionnaire utilizing as 5-point scale ranging from 5="Without any difficulty" to 1="Unable to do".
Efficacy outcomes include changes in the range of motion of the wrist (ROM) | Through study completion, up to 3 years
  Ranges include:
  0-75 degrees flexion 0-70 degrees extension 50 degrees radioulnar deviation arc
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the ankle using PROMIS 10 Global health | Through study completion, up to 3 years
  The PROMIS® is a set of participant-centered measures that evaluates and monitors the physical, mental, and social health in adults. Although unknown in osteoarthritis, the PROMIS® 10 Global Heath Survey was developed by the National Institute of Health and validated across a variety of chronic conditions. Each efficacy measure will be analyzed separately while accounting for potential confounding factors in the model such as age, sex, BMI, severity of OA diagnosis, smoking status, and past treatments in targeted joint. The Bonferroni adjustment for multiple testing correction will be used within each cohort. The PROMIS Global-10 is a 10-item patient-reported questionnaire utilizing as 5-point Global Physical Health Score scale ranging from 5="Excellent/Completely" to 1="Poor/Not at all" and a 5-point Global Mental Health scale ranging from 5="Never/None" to 1="Always/Very Severe", as well as a single 11-point question scale from 0="No Pain" to 10="Worst Pain Imaginable".
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the ankle using SF-12v2 | Through study completion, up to 3 years
  The SF-12v2 is a generic health outcome measurement widely used in chronic illness and chronic pain conditions. The SF-12v2 is a shorter tool that requires less patient and provider effort. Validity and feasibility have been reviewed with demonstration for significance in non-cancer pain patients. Each efficacy measure will be analyzed separately while accounting for potential confounding factors in the model such as age, sex, BMI, severity of OA diagnosis, smoking status, and past treatments in targeted joint. The Bonferroni adjustment for multiple testing correction will be used within each cohort. SF-12v2 patient-reported questionnaire is utilizes a 5-point scale ranging from "Excellent"/"All of the time" to "None of the time"/"Poor" for both physical and mental questions as well as a 3-point score ranging from "Yes, limited a lot" to "No, not limited at all" for two physical questions
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the ankle using the Pain Score on Visual Analog (VAS-Pain) | Through study completion, up to 3 years
  VAS instrument measures a characteristic that spans a continuum, cannot be precisely or optimally measured by or would lack sensitivity in distinguishing subtle changes on an ordinal scale. Pain intensity is a characteristic that is Sanford Health Confidential commonly measured in this manner. A 100-mm VAS will be administered to assess the subject's experience of joint pain intensity. Each efficacy measure will be analyzed separately while accounting for potential confounding factors in the model such as age, sex, BMI, severity of OA diagnosis, smoking status, and past treatments in targeted joint. The Bonferroni adjustment for multiple testing correction will be used within each cohort. The visual analog scale (VAS) patient-reported questionnaire is a subjective measure for acute and chronic pain utilizing a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain".
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the ankle using the Foot and Ankle Disability Index (FADI) | Through study completion, up to 3 years
  The Foot and Ankle Disability Index (FADI) is a 34-item questionnaire divided into two sub-scales: the Foot and Ankle Disability Index and the Foot and Ankle Sports Disability index (Hale 2005). Although not one foot and ankle self-reported measure has been determined as the most reliable, FADI is designed to detect deficits in higher functioning subjects and is more sensitive to responses after deliberate intervention. Each efficacy measure will be analyzed separately while accounting for potential confounding factors in the model such as age, sex, BMI, severity of OA diagnosis, smoking status, and past treatments in targeted joint. The Bonferroni adjustment for multiple testing correction will be used within each cohort. The FADI is a 34-item patient-reported questionnaire utilizing a 5-point scale ranging from 0% (most disability) to 100% (least disability), e.g. 0="Unable to do"/"Unbearable" to 4="No difficulty"/"No Pain".
Efficacy outcomes include changes in the range of motion of the ankle (ROM) | Through study completion, up to 3 years
  Ranges include:
  0-40 degrees plantar flexion 0-20 degrees dorsiflexion 0-30 degrees inversion 0-20 degrees eversion
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the hip using PROMIS 10 Global health | Through study completion, up to 3 years
  The PROMIS® is a set of participant-centered measures that evaluates and monitors the physical, mental, and social health in adults. Although unknown in osteoarthritis, the PROMIS® 10 Global Heath Survey was developed by the National Institute of Health and validated across a variety of chronic conditions. Each efficacy measure will be analyzed separately while accounting for potential confounding factors in the model such as age, sex, BMI, severity of OA diagnosis, smoking status, and past treatments in targeted joint. The Bonferroni adjustment for multiple testing correction will be used within each cohort. The PROMIS Global-10 is a 10-item patient-reported questionnaire utilizing as 5-point Global Physical Health Score scale ranging from 5="Excellent/Completely" to 1="Poor/Not at all" and a 5-point Global Mental Health scale ranging from 5="Never/None" to 1="Always/Very Severe", as well as a single 11-point question scale from 0="No Pain" to 10="Worst Pain Imaginable".
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the hip using SF-12v2 | Through study completion, up to 3 years
  The SF-12v2 is a generic health outcome measurement widely used. The Bonferroni adjustment for multiple testing correction will be used within each cohort. SF-12v2 patient-reported questionnaire is utilizes a 5-point scale ranging from "Excellent"/"All of the time" to "None of the time"/"Poor" for both physical and mental questions as well as a 3-point score ranging from "Yes, limited a lot" to "No, not limited at all" for two physical questions. The PROMIS Global-10 is a 10-item patient-reported questionnaire utilizing as 5-point Global Physical Health Score scale ranging from 5="Excellent/Completely" to 1="Poor/Not at all" and a 5-point Global Mental Health scale ranging from 5="Never/None" to 1="Always/Very Severe", as well as a single 11-point question scale from 0="No Pain" to 10="Worst Pain Imaginable".
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the hip using Pain Score on Visual Analog Scale (VAS-Pain) | Through study completion, up to 3 years
  A VAS instrument measures a characteristic that spans a continuum, cannot be precisely or optimally measured by or would lack sensitivity in distinguishing subtle changes on an ordinal scale. Pain intensity is a characteristic that is commonly measured in this manner. A 100-mm VAS will be administered to assess the subject's experience of joint pain intensity. Each efficacy measure will be analyzed separately while accounting for potential confounding factors in the model such as age, sex, BMI, severity of OA diagnosis, smoking status, and past treatments in targeted joint. The Bonferroni adjustment for multiple testing correction will be used within each cohort. The visual analog scale (VAS) patient-reported questionnaire is a subjective measure for acute and chronic pain utilizing a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain".
Efficacy outcomes include changes in patient reported outcomes (PRO) measurements for the hip using the Hip Disability Osteoarthritis Outcome Score (HOOS) | Through study completion, up to 3 years
  The HOOS is a patient-administered questionnaire consisting of 40 items across five subscales: Pain (10 items), Symptoms (5 items), Activity of Daily Living (17 items), Sport and Recreation Function (4 items) and Hip Related Quality of Life (4 items). The HOOS is scored on a Likert scale of 0 to 4 (no, mild, moderate, severe and extreme) with a total score is calculated by using a worst to best scale from 0 to 100, with 100 indicating no symptoms and 0 indicating extreme symptoms, with higher scores representing better function.
Efficacy outcomes include changes in the range of motion of the knee (ROM) measurements for the hip | Through study completion, up to 3 years
  Ranges include:
  0-125 degrees flexion 115-0 degrees extension 0-15 degrees hyperextension 0-45 degrees abduction 0-20 degrees adduction

SECONDARY OUTCOMES:
The secondary objective is to create a data registry for future research on ADRC use for OA | Through study completion, up to 3 years
  The registry will only contain treated individuals. Future analyses will analyze all subjects, subsets of subjects based on area of treatment, or potentially match treated subjects to similar control subjects for comparison of outcomes.

OTHER OUTCOMES:
A small volume of each subject's ADRC will be processed and stored for future research. | Through study completion, up to 3 years
  A small volume of each subject's ADRC will be processed and stored for future research.

CONTACTS AND LOCATIONS:
Overall Officials: David A. Pearce, PhD, Principal Investigator — Sanford Health
Locations (1):
- Sanford Orthopedics and Sports Medicine, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No